CLINICAL TRIAL: NCT03410498
Title: The Orthotic Effect of Functional Electrical Stimulation to Treat Foot Drop in People With MS Under Walking Conditions Simulating Those in Daily Life
Brief Title: The Effects of FES in a Variety of Walking Conditions in People With MS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen Margaret University (Other)
Responsible Party: Principal Investigator, Georgia Andreopoulou, Principal Investigator, Queen Margaret University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: QueenMU 12.1.2018
Record Dates: First submitted 2018-01-17; First posted 2018-01-25 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Stroop Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MS group (Other): This group will perform walking trials in various conditions, i.e. normal walking, walking whilst performing an attention demanding task and walking while being physically tired.
  Interventions: Other: Incremental shuttle walk test

INTERVENTIONS:
Other: Incremental shuttle walk test — In the incremental shuttle walk test, participants will have to walk between two cones (10m distance) several times. The time they will have to cover the distance between the two cones (signified by 'bleeps') will become increasingly shorter, until they cannot get to the next cone before the next 'bleep'. This test will last a maximum of 20 minutes.
  In the Stroop test, the words of four colours, but written with a different colour, will be projected on the wall in front of participants and they will need to identify the colour of the text and ignore the word itself.
  Other Names: Stroop test

SUMMARY:
The aim of this study is to measure the difference in the walking performance when functional electrical stimulation (FES) is on and off in people with MS that present foot drop under different 'real life' conditions, i.e. walking while doing another task that requires your attention and after been physically tired

DETAILED DESCRIPTION:
People with Multiple Sclerosis (pwMS) often experience foot drop, which means that the foot is not adequately lifted from the ground when walking. Functional Electrical Stimulation (FES) is applied to the shin muscles to aid lifting the foot of the ground and reduces the risk of trips and falls. PwMS that are users of functional electrical stimulation (FES) report that one of the benefits is that it reduces the mental effort of walking and that as a result less concentration is needed when they walk. Motor fatigability, which is the reduced ability of the muscles to produce force or power, also negatively affects the walking performance of pwMS. There have been several studies showing the benefits of FES to the walking of pwMS, but not while performing two tasks at the same time and experiencing fatigability resembling more daily life conditions. The proposed study aims to investigate the direct orthotic effect of FES (FES on vs off) in three different conditions, which include just walking, walking while performing an attention-demanding task and walking with an attention-demanding task after having completed a fatiguing task. The study design of this research allows the quantification of benefits of the use of FES which have until now only be reported subjectively.

ELIGIBILITY:
Inclusion Criteria:

For people with MS:

* Clinically definite multiple sclerosis according to the revised McDonald criteria.
* People with EDSS ≤ 5.0.
* People with MS who experience foot drop.
* Able to walk at least 200 meters unassisted, i.e without walking aids.

For healthy participants:

* Not been diagnosed with any neurological disease or have any other condition or injury which will affect walking ability.

Exclusion Criteria:

For people with MS:

* Clinically diagnosed relapse within the last month.
* Any musculoskeletal impairment that can affect walking ability.
* Cognitive impairments; with a score in the Multiple Sclerosis Neuropsychological Screening Questionnaire (MSNQ) ≤ 75.
* Depression and anxiety; with a score in Hospital Anxiety & Depression Scale (HADS) > 10.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2024-12-29 (Estimated); Study Completion 2024-12-29 (Estimated)

PRIMARY OUTCOMES:
3D gait analysis | Baseline
  The orthotic effect, i.e. the difference in ankle angle with the FES on and off.

SECONDARY OUTCOMES:
Stroop test/3D gait analysis | Baseline
  Dual task cost of walking speed

CONTACTS AND LOCATIONS:
Overall Officials: Thomas H Mercer, Prof., Study Chair — Queen Margaret University
Locations (1):
- Queen Margeret University, Musselburgh, United Kingdom